CLINICAL TRIAL: NCT00291057
Title: Phase II, Multi-center, Open-Label, Safety and Tolerance Study of a Novel Malathion Formulation in Infants and Toddlers With Pediculosis Capitis
Brief Title: Safety and Tolerability of a Novel Malathion Formulation in Infants and Toddlers With Head Lice
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Medical Director, Taro Pharmaceuticals USA
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MALG-0508
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-11

CONDITIONS: Lice Infestations
Keywords: Pediculosis; Head Lice
MeSH Terms: conditions — Lice Infestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): MALG
  Interventions: Drug: MALG

INTERVENTIONS:
Drug: MALG — 30 minute application

SUMMARY:
In a previous phase II study, the safety and efficacy of a novel formulation of malathion 0.5% was evaluated in patients 2 years of age and older. Based on the results of that study, this formulation is currently in a phase III study for that population.

The current study will use blood markers and clinical evaluations to determine the safety and tolerability of this formulation when used in children 6-24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed active head lice infestation
* Parent or guardian must be able to apply treatment

Exclusion Criteria:

* Allergy to pediculicides or hair care products
* Scalp conditions other than head lice
* Previous head lice treatment within the past 4 weeks
* Current antibiotic treatment

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2006-02; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in cholinesterase level | 1 day

SECONDARY OUTCOMES:
Clinical evidence of cholinesterase inhibition | 1 day
Local tolerability | 1 day
Cure of head lice 14 days after last treatment | 2 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Investigator Site, Scottsdale, Arizona
  - Investigator Site, St. Petersburg, Florida
  - Investigator Site, West Palm Beach, Florida
  - Investigator Site, New York, New York
  - Investigator Site, Miamiville, Ohio